CLINICAL TRIAL: NCT06517420
Title: The Effect of Kefir on Symptom Management and Quality of Life in Oncology Patients Treated With Chemotherapy
Brief Title: Effect of Kefir on Symptom Management and Quality of Life in Oncology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Aslıhan ÖZTÜRK ÇETİN, Research Assistant, Izmir Bakircay University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: BU-SBF-AÖC-01
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer; Colorectal Cancer
Keywords: kefir; symptom management; quality of life; chemotheraphy; oncology
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: A randomized controlled prospective experimental study
Who Masked: Participant, Outcomes Assessor
Masking Description: Simple random sampling method was used to avoid bias in providing patients to be included in the study before the data collection phase. With the computer-based randomization method, patients were numbered in the order of arrival and divided into experimental and control. The study data will be analyzed by an independent statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No intervention group) (No Intervention): Patients were asked "Individual Information Form, Nightingale Symptom Assessment Scale, FACT-G Quality of Life Scale, WHO Mucositis Evaluation Form, Rhodes Nausea Vomiting Gagging Index, ASCO Diarrhea Assessment Scale and Constipation Assessment Scale (CAS)" were filled in.
  No treatment was performed on the patients in the control group, and the patients continued their chemotherapy treatment.
  After 4 sessions, Nightingale Symptom Assessment Scale, FACT-G Quality of Life Scale, WHO Mucositis Evaluation Form, Rhodes Nausea Vomiting Gagging Index, ASCO Diarrhea Evaluation Scale and Constipation Assessment Scale (CAS)" were filled in again.
- Experimental group (intervention group) (Experimental): Patients were asked "Individual Information Form, Nightingale Symptom Assessment Scale, FACT-G Quality of Life Scale , WHO Mucositis Evaluation Form, Rhodes Nausea Vomiting Gagging Index, ASCO Diarrhea Assessment Scale and Constipation Assessment Scale (CAS)" were filled in.
  He was informed to consume 250 ml of kefir twice a day, before and after meals, for 1 week after the chemotherapy session, and to gargle in the mouth while consuming kefir, hold it for a while, and then swallow.
  At the end of each chemotherapy session and the 4th session, the Nightingale Symptom Assessment Scale, FACT-G Quality of Life Scale, WHO Mucositis Evaluation Form, Rhodes Nausea Vomiting Gagging Index, ASCO Diarrhea Assessment Scale and Constipation Assessment Scale (CAS) were applied by the practitioner. .
  Interventions: Other: kefir consumption

INTERVENTIONS:
Other: kefir consumption — Support and information was received from the Food Technology Department of a university's Experimental Medicine Application and Research Center. It was decided to choose the kefir to be used, which is produced from pasteurized cow's milk, lactase enzyme, probiotic culture (B. Lactis) and kefir culture, will meet the B12 need, contribute to increasing vitality and energy, and has the most suitable content in the market. Kefir, supplied by the researcher, was given to the patients at the end of each session in the amount that the patients should consume for a week, following the cold chain rule. While consuming kefir, it was recommended to gargle it in the mouth, hold it for a while, and then swallow. Patients were contacted for a week after the session to ensure that they applied kefir correctly.
  Arms: Experimental group (intervention group)

SUMMARY:
This study was planned as a randomized controlled prospective experimental study to determine the effect of kefir on symptom management and quality of life in oncology patients receiving chemotherapy. The population of the study consisted of 600 cancer patients who received chemotherapy in the outpatient chemotherapy unit of a university hospital between June 1, 2023 and February 1, 2024.

G*Power 3.1 package program was used to determine the number of samples. The sample size to ensure the power of the test (1-β = 0.80) was determined as a minimum of 26 people for each group. Considering the possibility of losses, 106 patients were included in the study. Data from 22 patients who were followed up during the preparation phase of the study were not included in the study. Simple random sampling method was used to avoid bias in providing patients to be included in the study before the data collection phase. With the computer-based randomization method, patients were numbered in the order of arrival and divided into experimental and control. The sample of the study was determined as 84, 42 in the experimental group and 42 in the control group.

In collecting data, "Individual Information Form, Nightingale Symptom Assessment Scale (NSD-S), FACT-G Quality of Life Scale, WHO Mucositis Evaluation Form, Rhodes Nausea Vomiting Gagging Index, ASCO Diarrhea Assessment Scale and Constipation Assessment Scale" were used. CAS)" was used.

DETAILED DESCRIPTION:
This study was planned as a randomized controlled prospective experimental study to determine the effect of kefir on symptom management and quality of life in oncology patients receiving chemotherapy. The population of the study consisted of 600 cancer patients who received chemotherapy in the outpatient chemotherapy unit of a university hospital between June 1, 2023 and February 1, 2024.

G*Power 3.1 package program was used to determine the number of samples. The sample size to ensure the power of the test (1-β = 0.80) was determined as a minimum of 26 people for each group. Considering the possibility of losses, 106 patients were included in the study. Data from 22 patients who were followed up during the preparation phase of the study were not included in the study. Simple random sampling method was used to avoid bias in providing patients to be included in the study before the data collection phase. With the computer-based randomization method, patients were numbered in the order of arrival and divided into experimental and control. The sample of the study was determined as 84, 42 in the experimental group and 42 in the control group.

In collecting data, "Individual Information Form, Nightingale Symptom Assessment Scale (NSD-S), FACT-G Quality of Life Scale, WHO Mucositis Evaluation Form, Rhodes Nausea Vomiting Gagging Index, ASCO Diarrhea Assessment Scale and Constipation Assessment Scale" were used. CAS)" was used.

Kefir, which is among the complementary treatments today, is a practice in the literature due to its positive effects in the management of many symptoms.

The use of kefir stands out because it can be applied regardless of place and time, is safe and cost-effective.

It is thought that kefir consumption, which has positive effects on many symptoms and strengthening the immune system, can be applied in the management of oral mucositis, nausea-vomiting, diarrhea and constipation, but the literature remains limited on this subject.

Since cancer patients, whose prevalence is increasing day by day, frequently experience symptoms during their treatment process, especially due to the chemotherapy they have received or are currently receiving, this study will add innovation to nursing science and literature and guide new research by determining whether kefir use is effective in symptom management and quality of life in oncology patients undergoing chemotherapy. It will happen.

ELIGIBILITY:
Inclusion Criteria:

* Being literate
* A diagnosis of breast and colorectal cancer
* Aged 18 or over
* The ability to communicate effectively and without language difficulties
* No diagnosis of mental or psychiatric illness
* No hearing or visual impairment
* No use of kefir, milk or dairy products prior to and/or during the treatment period
* The capacity to use a telephone for counselling

Exclusion Criteria:

* Having lactose intolerance,
* Allergy to milk and dairy products,
* Hearing and visual impairment,
* Not volunteering to participate in the study,
* Having mental disability or perception problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Nightingale Symptom Assessment Scale | 4 months
  Nightingale Symptom Assessment Scale (N-SDS) is a symptom assessment scale developed by Can and Aydıner for cancer patients in 2009 (Can and Aydıner, 2011). The scale (N-SDS), consisting of a total of 38 items, has three subscales (Physical Well-Being, Social Well-Being and Psychological Well-Being). When used alone, each item in the scale can reflect the extent to which cancer patients who are planning to receive or are receiving chemotherapy are affected by the problems caused by the disease/treatment, as well as how their quality of life is. While evaluating the scores on this Likert-type scale, the patient's response to the items is scored as "0" if the answer is no, "1" if the answer is very little, "2" if it is very little, "3" if it is little. "4" if many, "4" if many. A high score indicates that patients are highly affected by problems arising from the disease/treatment.
FACT-G Quality of Life Scale | 4 months
  The FACIT Measurement System is health-related Quality of Life (HRQOL) surveys targeting the management of chronic diseases. In FACT-G, Çetiner et al. It has been translated into Turkish by and its reliability and validity have been proven (Çetiner et al. 2004). The 4th version of the FACT-G survey is a compilation of 27 items and the general questions are divided into four main groups (Physical well-being, Social life and family well-being, Functional well-being, Emotional well-being). For each item of the rating scale; 0 points are given for the item "Not at all", 1 point for the item "Very little", 2 points for the item "Somewhat", 3 points for the item "A lot", and 3 points for the item "A lot". "4 points are given. An increase in the score obtained from the scale indicates that the quality of life is high.

SECONDARY OUTCOMES:
World Health Organization Mucositis Evaluation Form | 4 months
  It is used in clinics to evaluate the oral mucosa and grade oral mucositis. Generally, the scale is recommended for use in identifying toxicities caused by cytotoxic agents. Anatomical changes related to the oral mucosa and the severity of mucositis are scored between 0 and 4 points. In this scoring, the oral mucosa of the patients is evaluated objectively (erythema, ulceration, etc.), subjectively (oral pain, etc.) and functionally (patient's ability to eat, etc.). If these scores are 0, it is considered as no oral mucositis, while a score of '1' indicates that it is mild, a score of '2' indicates that it is moderate, a score of '3' indicates that it is serious, and a score of '4' indicates that it is at a life-threatening level (Çakmak and Nural, 2020).
Rhodes Index of Nausea, Vomiting and Retching | 4 months
  "Nausea-Vomiting and Gagging Index" was developed by Rhodes and McDaniel in 1999, and its validity and reliability were tested by Rhodes and McDaniel. The alpha internal consistency coefficient of the index is 0.98, and the alpha internal consistency coefficients of the subgroups vary between 0.83 and 0.99 (Rhodes and McDaniel, 1999). The adaptation of BKÖI to Turkish society was made by Genç (2010). In the adaptation made by Genç (2010), the internal consistency coefficient was found to be 0.95, and the alpha internal consistency number for subgroups was found to be between 0.81-0.95. In scoring the "Nausea-Vomiting and Gagging Index", items 1, 3, 6 and 7 are reversed. In scoring, for each answer, 4 means the highest level of distress and 0 means the least distress. The patient's experience of nausea and vomiting on each of the 8 items is collected. 32 is the highest possible value and indicates the most severe symptom formation (Genç, 2010).
American Society of Clinical Oncology (ASCO) Diarrhea Rating Scale | 4 months
  This fact sheet was developed by the American Society of Clinical Oncology (ASCO, 2022). All rights reserved worldwide. No sponsor was involved in the development of the content. It is the responsibility of the treating physician or other healthcare provider to determine medication dosages and the best dose, based on the patient's independent experience and knowledge. ASCO assumes no liability for any injury or damage to persons or property arising from or relating to any use of the information document or any errors or omissions. The information in ASCO's patient education materials is not intended to be medical advice or a substitute for medical advice. Patients with health care questions should call or see their physician or other health care provider immediately and should not disregard professional medical advice or delay seeking it because of information encountered here (ASCO, 2020).
Constipation Evaluation Scale (CAS) | 4 months
  The Constipation Assessment Scale was developed by McMillan and Williams (1989) to evaluate the constipation problem experienced by cancer patients in the last week (McMillan and Williams 1989). The original language of the scale is English. . The scale consists of 8 items and a single sub-dimension. The scale is prepared according to the three-point Likert type (0=No problems, 1=There are some problems, 2=There are serious problems) and the minimum score is 0 and the maximum score is 16. The scale score shows that the constipation problem is increasing. The patient rates each constipation item on a three-point scale (no problem to severe problem). Total scores range from 0 (no constipation) to 16 (worst possible constipation). The cutoff score for constipation has not been reported (McMillan and Williams, 1989; Wickham, 2016).

CONTACTS AND LOCATIONS:
Overall Officials: Olçun Ümit ÜNAL, Assos. Prof., Study Chair — HSU-Izmir Tepecik Training and Research Hospital, Bornova Oncology Hospital
Locations (1):
- Health Sciences University Izmir Tepecik Training and Research Hospital, Bornova Oncology Hospital, Additional Service Building, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No